CLINICAL TRIAL: NCT07118436
Title: Liquid Biopsy as a Biomarker in Patients Treated With PSMA Radioligand Therapy
Brief Title: Liquid Biopsy Under PSMA Radioligand Therapy
Acronym: LOOPS
Status: Recruiting | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital Augsburg (Other); Technical University of Munich (Other); German Research Foundation (Other)
Responsible Party: Principal Investigator, Kerstin Michalski, PD Dr. Kerstin Michalski, Wuerzburg University Hospital
Other Study IDs: GZ: MI 3238/1-1
Record Dates: First submitted 2025-07-28; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer Metastatic Castration-Resistant; Prostate Cancer
Keywords: mCRPC; PSMA; radioligand therapy; liquid biopsy; cfDNA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Weeks
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prostate cancer is the second most common cause of cancer death in men worldwide. After exhausting guideline-compliant therapies or in accordance with the approval of 177Lu-PSMA-617 (Pluvicto®), patients with metastatic castration-resistant prostate cancer (mCRPC) can be offered radioligand therapy (RLT) that targets the prostate-specific membrane antigen (PSMA). Despite an initially high response rate to PSMA-RLT, the disease often progresses rapidly again. The underlying mechanisms are still poorly understood.

Liquid biopsy (LBx) involves the collection and analysis of body fluids, particularly blood. Its major advantage compared to a tissue sample is its non-invasive nature, allowing for multiple samplings, as well as the examination of more than just a single punctured lesion. Among other things, circulating tumor DNA (ctDNA) can be detected in the blood.

The aim of this study is to apply LBx before, during, and after PSMA-RLT in patients with mCRPC to determine prognostic factors before therapy and to assess the value of LBx in evaluating treatment response. Furthermore, LBx will be used to gather information on the course of potential tumor heterogeneities and to determine resistance mechanisms against PSMA-RLT.

To this end, patients receiving PSMA-RLT will be enrolled in the study at three sites (University Hospital Wuerzburg, University Hospital Augsburg, Klinikum rechts der Isar Munich). The evaluation of clinical and imaging parameters will be carried out centrally at the University Hospital Wuerzburg, while the analysis of LBx will be performed at the University Hospital Augsburg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mCRPC eligble for PSMA RLT
* In-lable use for PSMA RLT
* PSMA PET/CT not older than 8 weeks prior to first cycle of PSMA RLT
* One previous line of antiandrogen receptor pathway treatment and one previous line of taxan based therapy
* Age ≥ 18 years
* Written informed consent
* Sufficient knowledge of the German language or presence of a translator

Exclusion Criteria:

* Unwilling to adhere to study procedures
* Missing interdisciplinary tumor conference advise for PSMA RLT

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic castration-resistant prostate cancer undergoing PSMA radioligand therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of LBx (precisely ctDNA) before PSMA RLT | 16-18 weeks
  identification of responders (partial response and stable disease)/non-responders (progressive disease) after 2 cycles of PSMA RLT, time-to-event analysis that could provide insights into overall survival or progression-free survival based on ctDNA level
Comparison of response assessment using LBx with biochemical response (PSA) after 2 cycles of PSMA RLT | 16-18 weeks
Comparison of response assessment using LBx with imaging-based response (PSMA PET/CT) after 2 cycles of PSMA RLT | 16-18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Michalski, MD, Principal Investigator — University hospital Wuerzburg - Department of Nuclear Medince; Rainer Claus, Prof., Principal Investigator — University hospital Augsburg - Internal Medicine II
Locations (3):
- Germany (3):
  - University hospital Wuerzburg - Department of Nuclear Medicine, Augsburg
  - TUM Klinikum rechts der Isar - Department of Nuclear medicine, München
  - University hospital Wuerzburg - Department of Nuclear Medicine, Würzburg